CLINICAL TRIAL: NCT06716359
Title: Comparison of the Effects of Hydromorphone and Nalbuphine Patient Controlled Analgesia in Postoperative Pain After Cesarean Section
Status: Enrolling by invitation | Type: Observational
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xianwei Zhang，MD, Professor, Huazhong University of Science and Technology
Other Study IDs: Acute postoperative pain
Record Dates: First submitted 2024-11-21; First posted 2024-12-04 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2024-11

CONDITIONS: Postoperative Pain; Patiet Controlled Analgesia
Keywords: postoperative pain; Cesarean section surgery; Hydromorphone; Nalbuphine; Predictive Model; patiet controlled analgesia
MeSH Terms: conditions — Pain, Postoperative | interventions — Observation; Methods

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cesarean section surgery: Observational study
  Interventions: Other: Observational study without intervention

INTERVENTIONS:
Other: Observational study without intervention — Observational study without intervention

SUMMARY:
Cesarean section is an essential surgical procedure in obstetrics, which not only addresses dystocia and certain obstetric syndromes, ensuring the safety of the maternal participants, but also increases perinatal survival rates and can save the mother's life. However, the surgical trauma and uterine contractions resulting from cesarean delivery lead to severe pain, which can hinder the mother's postoperative recovery and negatively affect her mental health. Therefore, improving postoperative pain management and addressing issues such as depression and anxiety are crucial challenges in clinical practice today.

Patient-controlled intravenous analgesia (PCA) is widely used in postoperative pain management after cesarean section due to its ability to maintain the minimum effective drug concentration, minimal fluctuation in drug levels, ease of management, and no restriction on activity. However, research on the effects and adverse reactions of hydromorphone and nalbuphine for postoperative pain relief in cesarean section is limited.

In this study, the investigators aim to compare the effects of hydromorphone hydrochloride and nalbuphine in obstetric PCA and examine how various clinical factors influence pain outcomes and adverse reactions. Based on multivariate analysis, the investigators further aim to construct and validate a predictive model for poor analgesic outcomes. To develop more personalized strategies for postoperative pain management following cesarean section, more personalized guidance strategies for postoperative pain management following cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 20 to 50 years old;
* ASA grades I to III;
* Full term pregnancy and planned cesarean section with transverse incision in the lower segment of the uterus;
* Pregnant women who are willing to participate in this study and sign informed consent forms.

Exclusion Criteria:

* Have a history of dementia, mental illness, or any central nervous system disorder;
* Pregnant women who are addicted to alcohol and drugs;
* Difficulty in follow-up or poor patient compliance;
* Has taken other investigational drugs or participated in other clinical trials in the three months prior to being selected for the study;
* Serious complications occur during delivery;
* Unable to cooperate with the research for any reason.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women planning to undergo cesarean section surgery
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2025-05-20 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of pain after caesarean section | 2024-12-05-2025-05-30
  Assessment of chronic postoperative pain by Brief Pain Inventory from 0 to ten, The higher the score, the stronger the pain
Incidence of inadequate analgesia | 2024-12-05-2025-05-30
  Postoperative pain is represented by NRS score (0-10). The higher the NRS score, the more severe the pain. A NRS score of ≥ 4 is considered inadequate analgesia.

SECONDARY OUTCOMES:
Adverse effects of postoperative analgesia | 2024-12-05-2025-05-30
  Incidence and the risk factors of adverse effects of postoperative analgesia
Usage of patient controlled analgesia (PCA) | 2024-12-05-2025-05-30
  Assessment of PCA Press Count and PCA Consumption
Diclofenac sodium dosage | 2024-12-05-2025-05-30
  Diclofenac sodium dosage after caesarean section
Patient satisfaction | 2024-12-05-2025-05-30
  Assessment of patient satisfaction by score from 0 to ten, The higher the score, the more satisfied the patient.
Length of hospital stay | 2024-12-05-2025-05-30
  Assessment of the length of hospital stay

OTHER OUTCOMES:
Regression analysis of inadequate analgesia | 2024-12-05-2025-05-30
  Univariate and multivariate regression analysis of inadequate postoperative analgesia. Postoperative pain is represented by NRS score (0-10). The higher the NRS score, the more severe the pain. A NRS score of ≥ 4 is considered inadequate analgesia.
Acute postoperative pain predictive model | 2024-12-05-2025-05-30
  Development and validation of a predictive model for acute postoperative pain after cesarean section.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sharpe EE, Booth JL, Houle TT, Pan PH, Harris LC, Aschenbrenner CA, Eisenach JC. Recovery of physical activity after cesarean delivery and its relationship with pain. Pain. 2019 Oct;160(10):2350-2357. doi: 10.1097/j.pain.0000000000001628. PMID 31145215
- [Background] Zhang Y, Betran AP, Li X, Liu D, Yuan N, Shang L, Lin W, Tu S, Wang L, Wu X, Zhu T, Zhang Y, Lu Z, Zheng L, Gu C, Fang J, Liu Z, Ma L, Cai Z, Yang X, Li H, Zhang H, Zhao X, Yan L, Wang L, Sun X, Luo Q, Liu L, Zhu J, Qin W, Yao Q, Dong S, Yang Y, Cui Z, He Y, Feng X, He L, Zhang H, Zhang L, Wang X, Souza JP, Qi H, Duan T, Zhang J. What is an appropriate caesarean delivery rate for China: a multicentre survey. BJOG. 2022 Jan;129(1):138-147. doi: 10.1111/1471-0528.16951. Epub 2021 Oct 26. PMID 34559941
- [Background] Li HT, Luo S, Trasande L, Hellerstein S, Kang C, Li JX, Zhang Y, Liu JM, Blustein J. Geographic Variations and Temporal Trends in Cesarean Delivery Rates in China, 2008-2014. JAMA. 2017 Jan 3;317(1):69-76. doi: 10.1001/jama.2016.18663. PMID 28030701
- [Background] Lumbiganon P, Laopaiboon M, Gulmezoglu AM, Souza JP, Taneepanichskul S, Ruyan P, Attygalle DE, Shrestha N, Mori R, Nguyen DH, Hoang TB, Rathavy T, Chuyun K, Cheang K, Festin M, Udomprasertgul V, Germar MJ, Yanqiu G, Roy M, Carroli G, Ba-Thike K, Filatova E, Villar J; World Health Organization Global Survey on Maternal and Perinatal Health Research Group. Method of delivery and pregnancy outcomes in Asia: the WHO global survey on maternal and perinatal health 2007-08. Lancet. 2010 Feb 6;375(9713):490-9. doi: 10.1016/S0140-6736(09)61870-5. Epub 2010 Jan 11. PMID 20071021
- [Background] Klemetti R, Che X, Gao Y, Raven J, Wu Z, Tang S, Hemminki E. Cesarean section delivery among primiparous women in rural China: an emerging epidemic. Am J Obstet Gynecol. 2010 Jan;202(1):65.e1-6. doi: 10.1016/j.ajog.2009.08.032. Epub 2009 Oct 12. PMID 19819416